CLINICAL TRIAL: NCT06066892
Title: Accuracy Evaluation of Different "All on Four" Impression Techniques Using Plaster Jig
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Doaa Abd El-Razik El-Mowafy, Faculty of dentistry, Mansoura University, Mansoura University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14120219RP
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Implant Prosthodontics
MeSH Terms: interventions — Dental Impression Technique

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital impression (Experimental): Digital impression using intraoral scanner
  Interventions: Procedure: Impression techniques
- One stage open impression technique (Experimental): Splinting impression long transfer and open tray impression technique
  Interventions: Procedure: Impression techniques
- Two stage closed tray and open tray (Experimental): Primary impression with closed tray impression techniques then secondary impression by open tray technique
  Interventions: Procedure: Impression techniques

INTERVENTIONS:
Procedure: Impression techniques — 3 types of impression techniques for all on four

SUMMARY:
This study will be conducted to evaluate the accuracy of different implant impression techniques using plaster jig Participants will have three types of impression techniques

ELIGIBILITY:
Inclusion Criteria:

Non smokers Good oral hygiene Free from any signs of implant failure and requesting a fixed prosthesis

Exclusion Criteria:

* patients that have severe bone resorption or excessive interarch space

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2023-10-16 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of impression technique | 3 months
  By using plaster jig

CONTACTS AND LOCATIONS:
Locations (1):
- Doaa Mowafy, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No